CLINICAL TRIAL: NCT06095310
Title: Evaluation of New Computer Vision Methods to Characterize Depression Severity in Patients Hospitalized for Severe Depression.
Brief Title: Clinical and Objective Psychiatric Analyses in Severe Depression.
Acronym: CALYPSO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0366; 2022-A01160-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2023-07-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-01

CONDITIONS: Depression
Keywords: Psychiatry; prediction; depression; objective psychiatry; personalized treatments; evolution and prognosis; computer science; artificial intelligence; innovation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homogeneous groups (Experimental)
  Interventions: Behavioral: New computer vision methods

INTERVENTIONS:
Behavioral: New computer vision methods — Clinical interview: Hamilton scale using multi-modal sensors (cameras, audio, bracelet, fNIRS)

SUMMARY:
Participation in the CALYPSO project will be offered to all patients with severe depression hospitalized in the adult psychiatry department of Lille CHU.

An initial visit will provide a standardized clinical assessment with: a medical history and history of the disease, a standardized structured Hamilton scale interview (scale with a score from 0 to 21; the higher the score, the more severe the depression) to assess the severity of depression, and a search for the different features of severe depression (melancholic, psychotic, anxious, catatonic, seasonal) using DSM-5 criteria (list of criteria to be validated to determine the type of clinical features). When assessing the severity of depression using the Hamilton scale interview, the patient will be seated in an armchair 2 to 3 meters from a camera on a tripod, positioned behind the clinician and enabling the entire interview to be recorded and, in particular, several observable and measurable psychiatric signs and symptoms, known as objective markers. From the video will be extracted face landmark and pose parameter using state-of-the-art open source software (Mediapipe) to analyze patients' emotional facial expressions and spatial movements. Moreover, a microphone will be used to capture the audio synchronously with the video. Speech will be automatically transcoded using state-of-the-art Automatic Speech Recognition system (DeepSpeech) to enable analysis of voice-related parameters (voice timbre, prosody, sound intensity). A recording of physical activity (3-axis accelerometer sensor; 32 Hz) and emotional reactivity (heart rate in beats per minute 1Hz; electrodermal activity 4 Hz; skin temperature in degrees 4 Hz; Empatica© bracelet) and brain activity (cerebral blood flow change index 10Hz; pulse rate in bpm 10Hz; 3-axis acceleration and angular velocity of the head 10Hz via functional Near-Infrared Spectroscopy (fNIRS) using a HOT-2000 wearable headset) will also be offered to the patient to complete the assessment. The Hamilton scale interview and recording of objective markers will be carried out weekly during the patient's hospitalization in an examination room specifically equipped for the project, on the second floor of the Fontan Hospital, in the psychiatry department of the Lille University hospital.

Longitudinal follow-up will be carried out with assessments at 3, 6 and 12 months after hospital discharge, including the Hamilton scale interview and recording of objective markers (i.e., emotional facial expressions, spatial movements, voice timbre, prosody, sound intensity, physical activity, heart rate, electrodermal activity, skin temperature).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years of age
* with severe depression as defined by DSM-5 criteria hospitalized in the adult psychiatry department of Lille University Hospital.
* Socially insured
* Patient willing to comply with all study procedures and duration.

Exclusion Criteria:

* Refusal to participate after receiving clear and fair information about the study
* Pregnant or breast-feeding women
* Person deprived of liberty or under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Severity of depression and clinical characteristics. | The primary outcome is measured at the initial visit, then at assessments at 3, 6 and 12 months after hospital discharge.
  The severity of depression will be assessed with the interview on the Hamilton scale (a scale with a score from 0 to 21; the higher the score, the more severe the depression), and clinical features will be determined according to DSM-5 criteria (list of criteria to be validated to determine the type of clinical features).

SECONDARY OUTCOMES:
Objective markers of remission of depressive episode | The secondary outcome is measured at the initial visit, then at assessments at 3, 6 and 12 months after hospital discharge.
  The interviews will be filmed and recorded in order to collect objective markers of depression (i.e., emotional facial expressions, spatial movements, voice timbre, prosody, sound intensity, physical activity, heart rate, electrodermal activity, skin temperature).